CLINICAL TRIAL: NCT05342168
Title: Comparison of Histological Results Obtained From a Mesh Sponge (CytospongeTM) and Traditional Esophageal Mucosal Biopsies in Children and Adolescents With Eosinophilic Esophagitis
Brief Title: Comparison of Histology From a Mesh Sponge and Traditional Esophageal Biopsies in Children and Adolescents With EoE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Margaret Marcon, Associate Professor, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10000073082
Record Dates: First submitted 2021-03-25; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Eosinophilic Esophagitis
Keywords: cytosponge; esophageal biopsy; Histology
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Intervention Model Description: cross sectional study comparing to tissue sampling methods
Masking Description: Each sample type is read by a pathologist blinded to the traditional ly obtained biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Histology (Experimental): Specimen samples from the tradition pinch esophageal biopsy and the supernatant sample obtained from the mesh sponge (Cytosponge TM) will each be fixed and stained. The eosinophil count per high power field for the mesh sponge sample and the traditional biopsy sample will be compared for each subject.
  Interventions: Diagnostic Test: Using a swallowed expanding sponge (Cytosponge TM) to obtain sampling of the esophageal musosa

INTERVENTIONS:
Diagnostic Test: Using a swallowed expanding sponge (Cytosponge TM) to obtain sampling of the esophageal musosa — A gelatin capsule containing the collapsed mesh sponge is swallowed with an attached string fixed to the cheek. After 8 minutes the gelatin capsule will have dissolved and the expanded soft mesh sponge can be with drawn sampling the surface of the esophagus on the way out. The sponge then will be spun and the supernant fixed, processed and stained.
  Other Names: Cytosponge

SUMMARY:
The aim of the present study is determining the accuracy, safety and tolerance of the CytospongeTM (expandable sponge within a gelatin capsule attached to a string) relative to traditional upper endoscopy and esophageal biopsies in older children and adolescents with a diagnosis of Eosinophilic Esophagitis (EoE) to follow up on treatment changes. The findings from this study could help determine whether the CytospongeTM is a more cost-effective alternative to traditional upper endoscopy for histologic follow-up in children and adolescents with EoE.

DETAILED DESCRIPTION:
This is a cross-sectional study in pediatric subjects comparing histologic findings on esophageal biopsies obtained during upper GI endoscopies to histologic findings on tissue samples obtained through the use of the CytospongeTM in a group of paediatric patients with a diagnosis of EoE. Subjects will swallow the Cytosponge capsule (attached to a string) several hours prior to their scheduled endoscopy for treatment assessment. An esophageal sample will be obtained by withdrawing the expanded sponge thru the esophagus. This will be sent to pathology and fixed and stained. The subject will also undergo routine upper endoscopy under conscious sedation and follow up biopsies obtained as per routine standard of care to assess current treatment for EoE. There will be a blinded comparison between the biopsies and the Cytosponge sample by two pediatric pathologist with experience with EoE. Subjects and their caregivers will also be surveyed on their experience using the Cytosponge compared to having endoscopy.

This study has been performed in adults with Eosinophilic Esophagitis and found that the samples obtained with the Cytosponge was equivalent to the endoscopically obtained biopspes with out having to use endoscopy. Adult subjects also preferred the Sponge over having an endoscopy. The Cytosponge was shown to be safe and effected. Even larger adult trials in screening for esophageal cancer have shown the Cytosponge is safe and effective at sampling the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Previous histologic diagnosis of eosinophilic esophagitis (symptoms of esophageal dysfunction and at least 15 eosinophils per high-power field on esophageal biopsy and after a comprehensive assessment of non-EoE disorders that could cause or potentially contribute to esophageal eosinophilia).1
* Capable of swallowing a capsule 3 cm in length (trial with 3 cm jelly candy).
* 10 to 18 years of age.
* Male or female.
* Able to give assent or consent.
* Scheduled for an upper gastrointestinal endoscopy with biopsies on the same day to assess response to therapy and make decisions regarding further management.

Exclusion Criteria:

* Unable to swallow the capsule.
* Unable to give assent or consent.
* History of esophageal stricture on either upper gastrointestinal barium study or previous upper gastrointestinal endoscopy of food impaction that required removal.
* History of portal hypertension or esophageal varices.
* History of solid organ transplantation.
* Known bleeding diathesis.
* On anticoagulation therapy.
* Known platelet count less than normal for age.
* Pregnancy.
* Need for intubation during endoscopy.
* History of previous esophageal surgery.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Eosinophil count per high power field obtained from Cytosponge supernant and endoscopic esophageal biopsies will be compared | 1 week
  Comparison of histology by counting the number of eosinophilis seen per high power field results from supernatant sample obtained via mesh sponge withdrawal thru the esophagus to samples obtained by the gold standard traditional esophageal biopsy.

SECONDARY OUTCOMES:
Likert scale (10 point) evaluating patient and caregiver satisfaction | immediately following the endoscopy procedure
  Both patient and caregiver satisfaction will be assessed comparing the sponge method verses tradition upper will endoscopy with biopsy using a 10 point likert scale (1 to 10) with 10 being the better outcome.
Questionairre evaluating Patient and caregiver satisfaction | immediately following endoscopy procedure
  Both patient and caregiver satisfaction will be assessed comparing the sponge method verses tradition upper will endoscopy with biopsy using a satisfaction questionnaire.
Histology comparison of supernant obtained from sponge and esophageal pinch biopses | one week
  Supernant samples and esophageal biopsies will be fixed and stained and then reviewed by the study pathologist to compare findings

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Marcon, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Sickkids, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katzka DA, Geno DM, Ravi A, Smyrk TC, Lao-Sirieix P, Miremadi A, Debiram I, O'Donovan M, Kita H, Kephart GM, Kryzer LA, Camilleri M, Alexander JA, Fitzgerald RC. Accuracy, safety, and tolerability of tissue collection by Cytosponge vs endoscopy for evaluation of eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2015 Jan;13(1):77-83.e2. doi: 10.1016/j.cgh.2014.06.026. Epub 2014 Jul 3. PMID 24997328
- [Background] Katzka DA, Smyrk TC, Alexander JA, Geno DM, Beitia RA, Chang AO, Shaheen NJ, Fitzgerald RC, Dellon ES. Accuracy and Safety of the Cytosponge for Assessing Histologic Activity in Eosinophilic Esophagitis: A Two-Center Study. Am J Gastroenterol. 2017 Oct;112(10):1538-1544. doi: 10.1038/ajg.2017.244. Epub 2017 Aug 15. PMID 28809387
- [Background] Januszewicz W, Tan WK, Lehovsky K, Debiram-Beecham I, Nuckcheddy T, Moist S, Kadri S, di Pietro M, Boussioutas A, Shaheen NJ, Katzka DA, Dellon ES, Fitzgerald RC; BEST1 and BEST2 study investigators. Safety and Acceptability of Esophageal Cytosponge Cell Collection Device in a Pooled Analysis of Data From Individual Patients. Clin Gastroenterol Hepatol. 2019 Mar;17(4):647-656.e1. doi: 10.1016/j.cgh.2018.07.043. Epub 2018 Aug 9. PMID 30099104
- [Background] Benaglia T, Sharples LD, Fitzgerald RC, Lyratzopoulos G. Health benefits and cost effectiveness of endoscopic and nonendoscopic cytosponge screening for Barrett's esophagus. Gastroenterology. 2013 Jan;144(1):62-73.e6. doi: 10.1053/j.gastro.2012.09.060. Epub 2012 Oct 3. PMID 23041329
- [Background] Dellon ES, Liacouras CA, Molina-Infante J, Furuta GT, Spergel JM, Zevit N, Spechler SJ, Attwood SE, Straumann A, Aceves SS, Alexander JA, Atkins D, Arva NC, Blanchard C, Bonis PA, Book WM, Capocelli KE, Chehade M, Cheng E, Collins MH, Davis CM, Dias JA, Di Lorenzo C, Dohil R, Dupont C, Falk GW, Ferreira CT, Fox A, Gonsalves NP, Gupta SK, Katzka DA, Kinoshita Y, Menard-Katcher C, Kodroff E, Metz DC, Miehlke S, Muir AB, Mukkada VA, Murch S, Nurko S, Ohtsuka Y, Orel R, Papadopoulou A, Peterson KA, Philpott H, Putnam PE, Richter JE, Rosen R, Rothenberg ME, Schoepfer A, Scott MM, Shah N, Sheikh J, Souza RF, Strobel MJ, Talley NJ, Vaezi MF, Vandenplas Y, Vieira MC, Walker MM, Wechsler JB, Wershil BK, Wen T, Yang GY, Hirano I, Bredenoord AJ. Updated International Consensus Diagnostic Criteria for Eosinophilic Esophagitis: Proceedings of the AGREE Conference. Gastroenterology. 2018 Oct;155(4):1022-1033.e10. doi: 10.1053/j.gastro.2018.07.009. Epub 2018 Sep 6. PMID 30009819